CLINICAL TRIAL: NCT06403410
Title: Evaluation of the Effectiveness of Delirium Prevention Guideline Utilization for Intensive Care Patients
Brief Title: Delirium Prevention Guideline for Intensive Care Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Ogretim Uyesi Serpil Topcu, Assistant Professor, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Delirium Prevention Guideline
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Delirium; Nurse's Role
Keywords: delirium; non-pharmacologic; nursing intervention
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: randomized controlled quasi-experimental study
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will utilize single-blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): In the intervention group, initially, the Patient Identification Form, RASS, and Nu-DESC will be administered. The RASS and Nu-DESC forms will continue to be applied once a day throughout the patient's follow-up period in the intensive care unit, every 12 hours. Each intervention group patient randomized will receive the Delirium Prevention Guideline. The guideline includes standard practices used by intensive care nurses in patient monitoring. In addition to routine follow-ups, eye masks and earplugs will be applied to patients in the intervention group between 24:00 and 06:00. It is expected that the guideline will be used once every 24 hours, in the morning, to ensure standardization
  Interventions: Other: Delirium Prevention Guideline
- Control (No Intervention): Routine delirium monitoring conducted in the intensive care clinic will be performed for patients in this group. There is no standard form used for delirium in the unit where the study is conducted. At the beginning of data collection, the Control group patients will undergo the Patient Identification Form, RASS, and Nu-DESC (once every 12 hours). The RASS and Nu-DESC forms will continue to be applied once a day throughout the patient's follow-up period in the intensive care unit. Data collection will be terminated in case of delirium development in patients.

INTERVENTIONS:
Other: Delirium Prevention Guideline — Each intervention group patient randomized will receive the Delirium Prevention Guideline. The guideline is designed to be followed by nurses. However, collaboration with the physician is required for some aspects of the guideline (pain control, ordering/follow-up of laboratory tests, etc.). Support will be obtained from the intensive care physician, who is a member of the research team, for these steps. The guideline includes standard practices used by intensive care nurses in patient monitoring. In addition to routine follow-ups, eye masks and earplugs will be applied to patients in the intervention group between 24:00 and 06:00.
  Arms: Experimental

SUMMARY:
Delirium is a complication characterized by fluctuations in orientation, memory, thinking, or behavior, with sudden onset of these changes. Studies have shown that pharmacological agents are the most significant risk factors for delirium in intensive care units. In recent years, the impact of non-pharmacological interventions in preventing delirium development has started to be discussed.

DETAILED DESCRIPTION:
Delirium is a complication characterized by fluctuations in orientation, memory, thinking, or behavior, with a sudden onset of these changes. Increased mortality and prolonged hospital stay have been identified in patients diagnosed with delirium. Advanced age, underlying urinary or respiratory tract infection, and existing cognitive impairment increase the risk of delirium development. Studies have shown that pharmacological agents are the most significant risk factors for delirium in intensive care units. However, environmental factors such as sound, continuous light, odors, invasive and non-invasive interventions, sensory overload, lack of meaningful verbal and cognitive stimuli, social isolation, immobilization, sleep disorders, temperature, drafts, and absence of windows in the environment are also indicated to contribute to delirium development. The presence of tubes, urinary catheters, invasive procedures, mechanical ventilation, and retention in the patient also increases the risk. In treatment, early detection and prevention of risk factors are prioritized. In case of development, efforts are made to prevent delirium-related complications and reduce its duration through pharmacological and non-pharmacological interventions. However, although many studies have been conducted on the prevention of delirium development with numerous pharmacological agents, a clear conclusion has not yet been reached. Pharmacological agents are generally used to alleviate symptoms. In recent years, the impact of non-pharmacological interventions in preventing delirium development has started to be discussed. Non-pharmacological interventions used in delirium prevention, as published by the National Institute for Health and Care Excellence (NICE), are itemized as pain management, prevention of dehydration, early mobilization, infection control, regulation of medications, sleep hygiene, and patient orientation. NICE also emphasizes the necessity of using a validated tool for assessing delirium.

A meta-analysis study has been published examining non-pharmacological interventions aimed at reducing the incidence of delirium, with a total of 26 studies included. According to this study, the methods that reduce the incidence are, respectively; family involvement, exercise program, multiple interventions (occupational therapy, reorientation, sleep therapy, music, etc.), ensuring cerebral hemodynamics, arranging the physical environment, and applying a sedation protocol. When the studies are examined, it is seen that efforts focus on ensuring sleep hygiene, maintaining patient orientation, and eliminating factors in the physical environment that may disrupt patient comfort. Evidence suggests strategies such as optimizing the environment, controlling light and noise, grouping patient care activities, and taking appropriate measures to preserve patients' sleep cycles to promote sleep regulation in adult ICU patients (Evidence: +1C). In the literature, studies have been conducted on the use of earplugs to protect ICU patients from noise and using eye masks to reduce exposure to light to ensure sleep hygiene. Delirium prevention strategies to be implemented should be compatible with clinical workflow. The method to be used should be easily adapted by all team members and patient relatives, and should be encouraged for use in clinical protocol. Collaboration between physicians, nurses, and patient relatives is essential in preventing delirium development. The pharmacological dimension of preventive interventions can be carried out by physicians, while non-pharmacological interventions can be implemented through collaboration between nurses and patient relatives. In this study, we aimed to determine the effect of guideline usage and team collaboration on the frequency of delirium development.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above,
* Without motor, sensory, or hearing impairment,
* Able to communicate,
* Admitted to the intensive care unit within the first 24 hours of admission,
* Without chronic cerebral damage,
* Richmond Agitation Sedation Scale value between -1 and +1 at the beginning of the study,
* Nursing Delirium Screening Scale (Nu-DESC) score <2,
* No wounds or infections in the ears or eyes,
* Patients who have given consent to participate in the study.

Exclusion Criteria:

* Patients who receive sedation or require sedation during the data collection process, those who are unable to communicate due to intubation, those with diagnosed psychiatric disorders, those with profound hearing loss affecting communication, and those who do not wish to use eye masks and earplugs will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
In patients receiving Delirium Prevention Guidelines, the rate of delirium development is change compared to the control group at the end of one week. | 3 weeks
  prevent delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Demiroğlu Bilim University, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researchers may share IPD data after the completion and publication of the study.

REFERENCES:
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the Intensive Care Unit: executive summary. Am J Health Syst Pharm. 2013 Jan 1;70(1):53-8. doi: 10.1093/ajhp/70.1.53. PMID 23261901
- [Background] Christensen M. What knowledge do ICU nurses have with regard to the effects of noise exposure in the Intensive Care Unit? Intensive Crit Care Nurs. 2005 Aug;21(4):199-207. doi: 10.1016/j.iccn.2005.01.003. Epub 2005 Feb 25. PMID 16039957
- [Background] Cinar F, Eti Aslan F. Evaluation of Postoperative Delirium: Validity and Reliability of the Nursing Delirium Screening Scale in the Turkish Language. Dement Geriatr Cogn Dis Extra. 2019 Dec 5;9(3):362-373. doi: 10.1159/000501903. eCollection 2019 Sep-Dec. PMID 31911787
- [Background] Deng LX, Cao L, Zhang LN, Peng XB, Zhang L. Non-pharmacological interventions to reduce the incidence and duration of delirium in critically ill patients: A systematic review and network meta-analysis. J Crit Care. 2020 Dec;60:241-248. doi: 10.1016/j.jcrc.2020.08.019. Epub 2020 Aug 31. PMID 32919363
- [Background] Duning T, Ilting-Reuke K, Beckhuis M, Oswald D. Postoperative delirium - treatment and prevention. Curr Opin Anaesthesiol. 2021 Feb 1;34(1):27-32. doi: 10.1097/ACO.0000000000000939. PMID 33315641
- [Background] Gaudreau JD, Gagnon P, Harel F, Tremblay A, Roy MA. Fast, systematic, and continuous delirium assessment in hospitalized patients: the nursing delirium screening scale. J Pain Symptom Manage. 2005 Apr;29(4):368-75. doi: 10.1016/j.jpainsymman.2004.07.009. PMID 15857740
- [Background] Litton E, Carnegie V, Elliott R, Webb SA. The Efficacy of Earplugs as a Sleep Hygiene Strategy for Reducing Delirium in the ICU: A Systematic Review and Meta-Analysis. Crit Care Med. 2016 May;44(5):992-9. doi: 10.1097/CCM.0000000000001557. PMID 26741578
- [Background] McManus J, Pathansali R, Stewart R, Macdonald A, Jackson S. Delirium post-stroke. Age Ageing. 2007 Nov;36(6):613-8. doi: 10.1093/ageing/afm140. Epub 2007 Oct 25. PMID 17965033
- [Background] McGuire BE, Basten CJ, Ryan CJ, Gallagher J. Intensive care unit syndrome: a dangerous misnomer. Arch Intern Med. 2000 Apr 10;160(7):906-9. doi: 10.1001/archinte.160.7.906. PMID 10761954
- [Background] Morandi A, Jackson JC, Ely EW. Delirium in the intensive care unit. Int Rev Psychiatry. 2009 Feb;21(1):43-58. doi: 10.1080/09540260802675296. PMID 19219712
- [Background] Delirium: prevention, diagnosis and management in hospital and long-term care. London: National Institute for Health and Care Excellence (NICE); 2023 Jan 18. Available from http://www.ncbi.nlm.nih.gov/books/NBK553009/ PMID 31971702
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Shi Q, Presutti R, Selchen D, Saposnik G. Delirium in acute stroke: a systematic review and meta-analysis. Stroke. 2012 Mar;43(3):645-9. doi: 10.1161/STROKEAHA.111.643726. Epub 2012 Jan 19. PMID 22267831
- [Background] Van Rompaey B, Elseviers MM, Van Drom W, Fromont V, Jorens PG. The effect of earplugs during the night on the onset of delirium and sleep perception: a randomized controlled trial in intensive care patients. Crit Care. 2012 May 4;16(3):R73. doi: 10.1186/cc11330. PMID 22559080